CLINICAL TRIAL: NCT06605066
Title: Post-Operative Physical Activity Monitoring: Algorithm Performance and Clinical Outcomes
Status: Completed | Type: Observational
Sponsor: Alp Ozel (Other)
Collaborators: Analog Device, Inc. (Other)
Responsible Party: Sponsor-Investigator, Alp Ozel, Assistant Professor, Abant Izzet Baysal University
Organization: Abant Izzet Baysal University (Other)
Other Study IDs: AIBU-FTR-AO-02
Record Dates: First submitted 2024-09-13; First posted 2024-09-20 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Postoperative Period; Physical Activity; Wearable Electronic Devices; Algorithms; Thoracic Surgery; Cardiac Surgery
Keywords: Postoperative Period; Physical Activity; Wearable Electronic Devices; Algorithms; Thoracic Surgery; Cardiac Surgery
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Post-Operative: Adults aged 18 and over who have undergone cardiac or thoracic surgery, been discharged from the post-anesthesia care unit, and transferred to an inpatient setting within 3 days prior to the data collection date.

SUMMARY:
The goal of this observational study is to validate physical activity algorithms in post-operative populations through raw accelerometer data collection using the ADI Study Watch 4.5 while in an in-patient setting. The secondary objective of the study is to collect skin temperature, photoplethysmography [PPG], Bioimpedance Analysis [BIA], heart rate [HR], SpO2, and electrodermal activity [EDA] using the ADI Study Watch 4.5. The main questions it aims to answer are:

* Can a wearable physical activity monitoring device assess patients' activity levels with higher accuracy and precision compared to traditional physical activity monitoring methods during the post-operative period?
* Do wearable devices placed on different body regions perform similarly in tracking physical activity during the post-operative period?
* Do post-operative physical activity monitoring algorithms improve patient compliance, accelerate recovery, and reduce hospital stay duration?
* Analysis of the activity tracking performance of a consumer device (Apple Watch) in patients after cardiac and thoracic surgery.

DETAILED DESCRIPTION:
Participants After obtaining ethical approval, individuals meeting the inclusion criteria will be enrolled in the study at BAİBÜ Izzet Baysal Training and Research Hospital. After providing participants with information about the study, they will be asked to sign an informed consent form. The total sample size for the preliminary t-test analysis was determined to be 42 with an alpha of 0.05, a power of 0.80, and a medium effect size using the G*Power (ver. 3.1.9.7) program. Anticipating a 40% drop-out rate, 60 individuals will be included in the study. To determine the final sample size, a power analysis will be performed using data obtained from the study.

Assessment Methods The demographic information of the participants will be collected using the Participant Identification Form. Pre-operative physical condition will be evaluated with the ASA Physical Status Classification System, skin color with the Fitzpatrick Skin Type Scale, pain level while resting, coughing, and moving will be assessed using the Visual Analog Scale (VAS), fatigue and anxiety with VAS, functional walking capacity with the 6-Minute Walk Test, physical activity level with the International Physical Activity Questionnaire, fear of movement with the TAMPA Scale of Kinesiophobia, and quality of life with the SF-36 Short Form.

The evaluation forms applied to the participants consist of the following sections:

1. Participant Identification Form 2. ASA Score 3. Fitzpatrick Skin Type Scale 4. Symptoms VAS (0-10) 5. Six-Minute Walk Test 6. International Physical Activity Questionnaire 7. TAMPA Scale of Kinesiophobia

1. Participant Identification Questions

   In the questionnaire, the following questions will be asked to determine the characteristics of the participants:

   Name-Surname, Gender, Date of Birth, Height, Weight Type of surgery, Arm length, Step length, Wrist circumference, Smoking: Participants will be asked whether they smoke, and the data will be recorded in pack-years. Educational level: After verbally asking participants about their educational level, it will be recorded as illiterate, primary school, middle school, high school, or university. Employment status: Participants' occupations will be asked verbally and recorded as housewife, employed, or retired. Medical history: Participants will be asked whether they have any chronic illnesses or have undergone surgery before. Medications: Participants will be asked whether they take any medications regularly, and the data will be recorded.
2. ASA Physical Status Classification System:

   The ASA system classifies patients' physical conditions before surgery as follows:

   ASA 1: A healthy and normal person with no disease or systemic disorder other than a surgical pathology that does not cause systemic dysfunction.

   ASA 2: A person with a systemic disorder caused by a surgical condition or a disease such as mild emphysema, chronic bronchitis, diabetes, hypertension, or anemia.

   ASA 3: A person with a disease that limits activity but is not incapacitating, such as heart failure, a previous myocardial infarction, hypovolemia, advanced diabetes, or limited lung function.

   ASA 4: A person with a disease, such as respiratory disease, kidney or liver failure, that severely impairs physical ability and poses a constant threat to life.

   ASA 5: A moribund person not expected to survive 24 hours without surgery. ASA 6: This group includes brain-dead patients who are suitable for organ donation.
3. Fitzpatrick Skin Type Scale:

   Participants' skin types will be categorized into six groups, from very fair (skin type I) to very dark (skin type VI), according to the Fitzpatrick Skin Type Scale, which is commonly used in the literature to determine skin type. Skin type is characterized by general appearance, eye color, hair type and color, etc.

   Type I - Very fair skin, sensitive to the sun, light eye color (blue/green), blonde or light brown hair.

   Type II - Fair skin, light brown or brown hair, light-colored eyes. Type III - Fair to wheatish skin, light or dark eyes, brown or black hair. Type IV - Wheatish skin, dark eyes (brown/black), brown or black hair. Type V - Dark brown skin, dark (black) eyes, black hair. Type VI - Very dark skin (almost black), black eyes, black hair.
4. Visual Analog Scale (VAS):

   Pain levels will be assessed using the VAS. According to the VAS, pain severity is generally rated on a 0-10 cm scale, with "no pain" being 0 and "the worst pain imaginable" being 10. Pain severity categories are:

   <3: mild pain, 3-6: moderate pain, 6: severe pain.
5. Six-Minute Walk Test (6MWT):

   As an easily applicable and objective assessment, the 6MWT is the most widely used cardiopulmonary exercise test. Participants are asked to walk the longest possible distance in a straight corridor marked at 30 meters during six minutes. Before and after the test, heart rate, blood pressure, and oxygen saturation (SpO2) will be measured; dyspnea will be recorded using the Modified Borg Scale. The distance walked in six minutes will be noted in meters. A distance of less than 300 meters is associated with higher mortality. The normal range for healthy individuals is between 500 and 700 meters. The expected 6MWT distance will be calculated using the following formulas:

   Male: (7.57 X heightcm) - (5.02 X age) - (1.76 X weightkg) - 309 Female: (2.11 X heightcm) - (2.29 X weightkg) - (5.78 X age) + 667
6. International Physical Activity Questionnaire (Short Form):

   Developed by Craig in 2003 to assess physical activity levels in adults, the reliability and validity of this questionnaire were tested by Sağlam et al. in 2010. It assesses the types of physical activity individuals have performed in the past seven days and the time spent on each activity. It consists of seven questions, and the total score is calculated by multiplying the duration (minutes) and frequency (days) of moderate and vigorous activities. Patients are classified as inactive (<600 MET min/week), moderately active (600-3000 MET min/week), or active (>3000 kcal/min).
7. TAMPA Scale of Kinesiophobia:

This is a 17-item self-report scale developed to measure fear of movement. Scores range from 17 to 68. Higher scores indicate greater fear of movement, while lower scores suggest minimal fear.

Participants who meet the inclusion criteria will wear the sensors for 5 hours after discharge from the ward. During this time, they are free to engage in natural activities. During data collection, the ADI Study Watch 4.5 will be worn on the left wrist, arm, and chest, the Apple Watch 8 will be worn on the right arm, and the Axivity AX6 on the ankle.

Statistics Descriptive statistics will be presented as mean and standard deviation for numerical variables or median and minimum-maximum values. Categorical variables will be described as numbers and percentages. The Shapiro-Wilk test will be used to assess normality. An independent t-test will be used to compare two groups when assumptions are met, and the Mann-Whitney U test will be used when assumptions are not met. Correlations between parameters will be examined using Spearman or Pearson correlation analysis, depending on normality. Chi-square tests will be used to examine differences between categorical variables. The significance level will be set at p<0.05. Data analysis will be performed using the Statistical Package for the Social Sciences (SPSS) v.20.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18, male or female
* ASA Score II - III
* Patients booked for a surgical procedure requiring general anesthesia care
* The subject has had a surgical procedure ≤3 days prior to data collection
* Expected duration of general anesthesia to be > 1 hour
* Expected to be transferred to the PACU from the operating room
* Patients with an expected duration in the PACU ≥ 45 minutes
* Expected to be transferred from the PACU to an in-patient setting
* Must be able to understand and provide written consent
* Must be willing and able to comply with study procedures and duration

Exclusion Criteria:

* The subject is unable or unwilling to provide written consent
* The subject is unable or unwilling to comply with the study and duration
* The subject has not yet recovered from the effects of anesthesia
* The subject requires the use of a wheel chair
* The subject has been diagnosed with a movement disorder such as Parkinson's disease, ataxia, dystonia, etc.
* The subject has not yet recovered from knee or hip surgery
* The subject has undergone orthopedic surgery within the last 2 years
* The subject has an injury, deformity, or abnormality at the sensor site that in the opinion of the investigators would interfere with the sensors' function
* The subject has any other condition, which in the opinion of the investigator would make them unsuitable for the study
* The subject is pregnant, lactating, or trying to get pregnant.
* Subjects with a history of severe contact allergies that may cause a reaction to standard adhesive materials found medical tape.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals who meet the inclusion criteria and have undergone Cardiovascular or Thoracic surgery at Izzet Baysal Training and Research Hospital will be included in the study. Individuals will be included in the study according to the simple random sampling method.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2024-10-09 (Actual); Primary Completion 2025-07-21 (Actual); Study Completion 2025-07-21 (Actual)

PRIMARY OUTCOMES:
Raw Accelerometer Data | Within 3 days after the patient is discharged to the inpatient setting, data will be collected from each individual once for a duration of 5 hours using wearable devices.
  Accelerometers measure linear acceleration (specified in mV/g) along one or several axis. ADI Study Watch 4.5 and Axivity AX6 devices have a three-axis accelerometer, which delivers acceleration values in each of the three axes. The values reported by the accelerometers are measured in increments of the gravitational acceleration, with the value 1.0 representing an acceleration of 9.8 meters per second (per second) in the given direction. Acceleration values may be positive or negative depending on the direction of the acceleration. Raw accelerometer data will be used to validate step count, distance and activity level algorithms. Measurements will be made with ADI Study Watch 4.5 and Axivity AX6.

SECONDARY OUTCOMES:
International Physical Activity Questionnaire (Short Form) | Once during the study period, within 3 days after the patient is discharged to the inpatient setting.
  The questionnaire can determine the type of physical activity individuals have done in the last seven days and the time they spent. It consists of a total of 7 questions. The total score is calculated by multiplying the duration (minutes) and frequency (days) of moderate and vigorous activity. Patients with a metabolic equivalent score of less than 600 MET min/week will be considered inactive, 600-3000 MET min/week will be considered moderately active, and patients with more than 3000 kcal/min will be considered active.
Six Minute Walk Test | Once during the study period, within 3 days after the patient is discharged to the inpatient setting.
  In this test, subjects are asked to reach the longest possible walking distance in six minutes on a 30-meter track marked in a straight corridor. Before and after the test, the individual&#39;s heart rate, blood pressure and oxygen saturation (SpO2) are measured; the degree of dyspnea is determined and recorded according to the Modified Borg scale. At the end of the test, the individual&#39;s six-minute walking distance is noted in meters. A distance walked in six minutes of less than 300 meters is associated with mortality. This distance varies in healthy individuals, but is between 500-700 meters. In studies conducted, equations have been developed to obtain reference values for 6MWT in healthy individuals. Expected 6MWT distances will be calculated according to the following formulas: Male: (7.57 X heightcm)- (5.02 X age)-(1.76 X kg)-309 Female: (2.11 X heightcm)- (2.29 X kg)- (5.78 X age)+ 667
Visual Analogue Scale (VAS) | Once during the study period, within 3 days after the patient is discharged to the inpatient setting.
  Pain intensity at rest, pain intensity when coughing, pain intensity when moving, fatigue severity, and anxiety state will be assessed by VAS. According to the VAS, pain severity is generally rated on a scale where no pain; is 0 points and the worst imaginable pain; is 10 points (on a 10 cm scale). The severity ranges are classified as follows: less than 3 is considered mild, between 3-6 is moderate, and greater than 6 is severe.
TAMPA Kinesiophobia Scale | Once during the study period, within 3 days after the patient is discharged to the inpatient setting.
  It is a self-reported 17-item scale developed to measure fear of movement. The lowest possible score is 17 and the highest is 68. A high score indicates a high level of fear of movement, while a low score indicates a negligible level of fear of movement.
ASA Physical Status Classification System | Once during the study period, within 3 days after the patient is discharged to the inpatient setting.
  The patient classification of ASA, which is an evaluation system in which patients are classified according to their physical condition before the operation, is as follows:
  ASA 1: A healthy and normal person who does not have any disease or any systemic disorder other than surgical pathology that does not cause a systemic disorder.
  ASA 2: A person who has a systemic disorder due to a cause requiring surgical operation or a disease such as low-level emphysema, chronic bronchitis, diabetes, hypertension, anemia, etc.
  ASA 3: A person who has a disease that limits their activity due to heart failure, previous myocardial infarction, hypovolemia, advanced diabetes, limited lung function, etc., but does not leave them weak.
  ASA 4: A person who has a disease such as respiratory system disease, kidney or liver failure, etc. that causes them to lose their strength completely and poses a constant threat to their life.
  ASA 5: A person who is expected to live no more than 24 hours and is in a stat
Bioimpedance Analysis | Within 3 days after the patient is discharged to the ward, data will be collected from each individual once for a duration of 5 hours using wearable devices.
  Bioimpedance analysis (BIA) is a method of estimating body fluid volumes by measuring the resistance to a high-frequency, low-amplitude alternating electric current. BIA, low cost and a commonly used approach for body composition measurements and assessment of clinical condition. ADI Study Watch 4.5 will be used to make the measurements.
Step Count | Within 3 days after the patient is discharged to the inpatient setting, data will be collected from each individual once for a duration of 5 hours using wearable devices.
  The number of steps will be calculated from the accelerometer and gyroscope information by making use of the built-in programmes on devices ADI Study Watch 4.5 and Axivity AX6. Step count measured by the Apple Watch Series 8 will be used for comparison.
Skin Temperature | Within 3 days after the patient is discharged to the inpatient setting, data will be collected from each individual once for a duration of 5 hours using wearable devices.
  Skin Temperature Sensors are specifically designed for continuous temperature monitoring using the skin as an indicator of body temperature. In contrast to the core body temperature, which is usually fairly constant around +37 degrees Celsius, the temperature of the skin can vary much more. A change in skin temperature of +-1 degree Celsius / +-1.8 degree Fahrenheit is considered usual. ADI Study Watch 4.5 will be used to make the measurements.
Electrodermal Activity | Within 3 days after the patient is discharged to the inpatient setting, data will be collected from each individual once for a duration of 5 hours using wearable devices.
  Electrodermal activity (EDA) is a measurement of eccrine activity that is influenced by sympathetic nervous system activity, resulting from environmental stimuli. EDA is an autonomic (involuntary) response. The physiological basis for EDA is neurological control of the rate of sweat gland production in the extremities, most notably the fingertips, palms of the hand, and soles of the feet. ADI Study Watch 4.5 is placed on the participant and a very low constant voltage applied (not felt by the participant). Then the current flowing as a result of this applied voltage is measured and converted to a conductance in accordance with Ohm's law. Skin conductance is measured in units of microsiemens, with normal human EDA ranging from 1 to 20 microsiemens.
Oxygen Saturation (SpO2) | Within 3 days after the patient is discharged to the ward, data will be collected from each individual once for a duration of 5 hours using wearable devices.
  ADI Study Watch 4.5 will be used to find out a persons oxygen saturation (SpO2) and analyse the readings using existing software. For most people, a normal pulse oximeter reading for your SpO2 level is between 95% and 100%.
Heart Rate Data | Within 3 days after the patient is discharged to the inpatient setting, data will be collected from each individual once for a duration of 5 hours using wearable devices.
  ADI Study Watch 4.5 will be used to find out a persons heart rate and analyse the readings using existing software. A normal resting heart rate for adults ranges from 60 to 100 beats per minute.
Gyroscope Data | Within 3 days after the patient is discharged to the inpatient setting, data will be collected from each individual once for a duration of 5 hours using wearable devices.
  A gyroscope measures angular velocity (specified in mV/deg/s). Measurements will be made with Axivity AX6.
Photoplethysmography Data | Within 3 days after the patient is discharged to the ward, data will be collected from each individual once for a duration of 5 hours using wearable devices.
  Photoplethysmography (PPG) is a simple optical technique used to detect volumetric changes in blood in peripheral circulation. It is a low cost and non-invasive method that makes measurements at the surface of the skin. PPG shows the blood flow changes as a waveform with the help of a bar or a graph. The waveform has an alternating current (AC) component and a direct current (DC) component. The AC component corresponds to variations in blood volume in syncronization with the heart beat. The DC component arises from the optical signals reflected or transmitted by the tissues and is determined by the tissue structure as well as venous and arterial blood volumes. The DC component shows minor changes with respiration. The basic frequency of the AC component varies with the heart rate and is superimposed on the DC baseline. ADI Study Watch 4.5 will be used to make the measurements.
Distance Traveled | Within 3 days after the patient is discharged to the ward, data will be collected from each individual once for a duration of 5 hours using wearable devices.
  Distance walked in metres will be calculated from accelerometer and gyroscope information using the built-in programs in the ADI Study Watch 4.5 and Axivity AX6. The distance measured by the Apple Watch Series 8 will be used for comparison.

CONTACTS AND LOCATIONS:
Locations (1):
- Bolu Abant Izzet Baysal University, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Since a commercial product will be developed, it is not yet clear which data will be shared.